CLINICAL TRIAL: NCT04272034
Title: A Phase 1 Study Exploring the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of INCB099318 in Participants With Select Advanced Solid Tumors
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of INCB099318 in Participants With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: A business decision was made to discontinue further enrollment. There were no safety concerns that contributed to this decision.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 99318-122; 2019-004990-21 (EudraCT Number)
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumors; MSI-H/dMMR Tumors; Cutaneous Squamous Cell Carcinoma; Urothelial Carcinoma, HCC; Cervical Cancer; Esophageal Squamous Cell Carcinoma; Merkel Cell Carcinoma; Small-cell Lung Cancer; Mesothelioma; PD-L1 Amplified Tumor (9p24.1); Nasopharyngeal Carcinoma; Cyclin-dependent Kinase 12 Mutated Tumors; Basal Cell Carcinoma (Unresectable or Metastatic); Sarcomatoid Renal Cell Carcinoma; Clear Cell Ovarian or Endometrial Carcinoma; Anal Carcinoma; Squamous Cell Penile Carcinoma; DNA Polymerase Epsilon Mutated Tumors (P286R and V411L)
Keywords: Advanced solid tumors
MeSH Terms: conditions — Carcinoma, Transitional Cell; Uterine Cervical Neoplasms; Esophageal Squamous Cell Carcinoma; Carcinoma, Merkel Cell; Small Cell Lung Carcinoma; Mesothelioma; Nasopharyngeal Carcinoma; Carcinoma, Basal Cell; Neoplasm Metastasis; Carcinoma, Renal Cell; Endometrial Neoplasms; Anus Neoplasms

STUDY DESIGN:
Intervention Model Description: The study consists of 2 parts. Part 1 is a dose-escalation design to identify the maximum tolerated dose and/or pharmacologically active dose for INCB099318. Part 2 is an expansion at 1 or more dose levels to further explore safety, preliminary efficacy, pharmacoketics, and pharmacodynamic effects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Participants with select solid tumors who are immunotherapy treatment-naive
  Interventions: Drug: INCB099318
- Cohort 2 (Experimental): Participants with high microsatellite instability (MSI-H) or deficient mismatch repair (dMMR) tumors who are immunotherapy treatment-naïve.
  Interventions: Drug: INCB099318
- Cohort 3 (Experimental): Participants with progression of any solid tumor treated with an approved anti-PD-1 monoclonal antibody therapy
  Interventions: Drug: INCB099318

INTERVENTIONS:
Drug: INCB099318 — INCB099318 administered orally in 20 mg or 100 mg tablets once daily or twice daily on each day of each 28-day cycle.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability, pharmacokinetics, and pharmacodynamics of INCB099318 in select solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Must have disease progression after treatment with available therapies that are known to confer clinical benefit or must be intolerant to or ineligible for standard treatment.
* Histologically confirmed advanced solid tumors (protocol-defined select solid tumors) with measurable lesions per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1) that are considered nonamenable to surgery or other curative treatments or procedures.
* ECOG performance status score of 0 or 1.
* Life expectancy > 12 weeks.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

Exclusion Criteria:

* Laboratory values outside the Protocol-defined ranges.
* Clinically significant cardiac disease.
* History or presence of an ECG that, in the investigator's opinion, is clinically meaningful.
* Untreated brain or central nervous system (CNS) metastases or brain or CNS metastases that have progressed (eg, evidence of new or enlarging brain metastasis or new neurological symptoms attributable to brain or CNS metastases).
* Known additional malignancy that is progressing or requires active treatment.
* Has not recovered to ≤ Grade 1 or baseline from toxic effects of prior therapy (including prior IO) and/or complications from prior surgical intervention before starting study treatment.
* Prior receipt of an anti-PD-L1 therapy.
* Treatment with anticancer medications or investigational drugs within protocol-defined intervals before the first administration of study drug.
* A 28-day washout for systemic antibiotics is required.
* Probiotic usage while on study and during screening is prohibited.
* Active infection requiring systemic therapy.
* Known history of HIV
* Evidence of hepatitis B virus or hepatitis C virus infection or risk of reactivation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events | Up to approximately 25 months
  Defined as any adverse event either reported for the first time or worsening of a pre-existing event after first dose of study drug up to 30 days after last dose of study drug.

SECONDARY OUTCOMES:
Cmax of INCB099318 | Up to approximately 3 months
  Maximum observed plasma concentration
tmax of INCB099318 | Up to approximately 3 months
  Time to maximum plasma concentration
Cmin of INCB099318 | Up to approximately 3 months
  Minimum observed plasma concentration over the dose interval
AUC0-t of INCB099318 | Up to approximately 3 months
  Area under the plasma concentration-time curve from time = 0 to the last measurable concentration at time = t
t½ of INCB099318 | Up to approximately 3 months
  Apparent terminal-phase disposition half-life
λz of INCB099318 | Up to approximately 3 months
  Terminal elimination rate constant
CL/F of INCB099318 | Up to approximately 3 months
  Oral dose clearance
Vz/F of INCB099318 | Up to approximately 3 months
  Apparent oral dose volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Louis Viviers, MD, Study Director — Incyte Corporation
Locations (24):
- United States (3):
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Prisma Health Cancer Institute Faris, Greenville, South Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
- Belgium (5):
  - Universitair Ziekenhuis Brussel, Brussels
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen (Uza), Edegem
  - Ghent University Hospital, Ghent
  - Universitaire Ziekenhuis Leuven - Gasthuisberg, Leuven
- Rigshospitalet Uni of Hospital of Copenhagen, Copenhagen, Denmark
- Finland (4):
  - Helsinki University Central Hospital, Helsinki
  - Docrates Cancer Center, Helsinki
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Karolinska University Hospital Solna, Solna
  - Uppsala Universitet - Akademiska Sjukhuset, Uppsala
- United Kingdom (6):
  - Western General Hospital, Edinburgh
  - St James University Hospital, Leeds
  - Guys and St Thomas Nhs Foundation Trust, London
  - The Royal Marsden Hospital Nhs Trust London, London
  - Imperial College Healthcare Nhs Trust - Hammersmith Hospital, London
  - Freeman Hospital Newcastle Upon Tyne Foundation Nhs Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No
Access to patient level data is not available for this study